CLINICAL TRIAL: NCT05793723
Title: Evaluation of Long-term Respiratory Complications in Infants With Perinatal COVID-19: a Pilot Study.
Brief Title: Long-term Respiratory Complications in Infants With Perinatal COVID-19
Acronym: COLF
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 4949
Record Dates: First submitted 2023-02-08; First posted 2023-03-31 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-03

CONDITIONS: COVID-19; Infant, Newborn, Diseases; Respiratory Function Tests
MeSH Terms: conditions — COVID-19; Infant, Newborn, Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Infants with confirmed neonatal COVID-19 infection
  Interventions: Diagnostic Test: Pulmonary function testing device
- Controls: Infants born to mothers with no history of COVID-19 infection during pregnancy and no neonatal COVID-19 infection
  Interventions: Diagnostic Test: Pulmonary function testing device

INTERVENTIONS:
Diagnostic Test: Pulmonary function testing device — Patients will undergo pulmonary function tests with the Exhalyzer D (Ecomedics, Switzerland) device. This device consists of 1) an ultrasonic flow measuring system for measuring flow, volume and molecular mass, 2) a nitrogen washout system to measure functional residual capacity (FRC) and other indices, 3) a carbon dioxide infrared measurement device for monitoring the level of carbon dioxide in exhaled breath.

SUMMARY:
Study outcomes and endpoints:

* Primary outcome: to assess clinical characteristics of infants with confirmed COVID-19 infection at birth and to evaluate long-term respiratory consequences of neonatal COVID-19 infection.
* Secondary outcome: to evaluate the prevalence and natural history of lung function impairment among infants with confirmed COVID-19 compared to infants with no history of COVID-19. To this end, infants will undergo pulmonary function testing (PFT) with the Exhalyzer D device (Eco Medics, Switzerland).

DETAILED DESCRIPTION:
In this prospective, observational longitudinal study, infants will undergo clinical and growth assessment at 6 and 12 months' follow-up. Respiratory complications, such as wheezing, infections, chronic cough will be recorded along with hospital admissions and drug prescription or use.

Infants will undergo PFT with the infants in the supine position, during quiet, natural sleep, according to American Thoracic Society/European Respiratory Society recommendations with measurement of lung volumes, flow, functional residual capacity, time to peak tidal expiratory flow/expiratory time ratio (tPTEF/tE)10. Lung ultrasound will be performed to rule out lung abnormalities. After allowing adaptation to the mask, the investigators will record tidal breathing, flow volume loops for >2 minutes or >20 artifact-free breaths. Using commercially available software (Spiroware, Ecomedics), the investigators will extract tidal breathing parameters: ratio of time to reach peak tidal expiratory flow to expiratory time (tPTEF/tE), tidal volume (VT), and respiratory rate (RR). tPTEF/tE is a reproducible and reliable marker of airway obstruction, can detect severe expiratory airway obstruction in infants with respiratory complaints and is associated with subsequent wheezing in infancy.

Appropriate statistical methods will be used to describe clinical characteristics of patients and compare groups (T-test, Mann-Whitney test, chi-squared test, multivariate analysis, mixed models depending on data distribution - evaluated with Shapiro-Wilk test - and data characteristics).

ELIGIBILITY:
Inclusion Criteria:

* term infants;
* informed consent;
* history of perinatal COVID-19 (confirmed by nasopharyngeal swab tests, study group)

Exclusion Criteria:

* congenital malformations (particularly airway malformations);
* lack of informed consent

Ages: 3 Months to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: In this prospective, observational longitudinal study, infants with and without history of COVID-19 will undergo clinical and growth assessment at 6 and 12 months' follow-up. Respiratory complications, such as wheezing, infections, chronic cough will be recorded along with hospital admissions and drug prescription or use. Pulmonary function tests will be performed during spontaneous, quiet sleep.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Clinical respiratory consequences of neonatal COVID-19 infection | 6 months of life
  Number or patients with wheezing, use of bronchodilators, steroids, hospitalizations for respiratory causes
Clinical respiratory consequences of neonatal COVID-19 infection (i.e. wheezing) | 12 months of life
  Number or patients with wheezing, use of bronchodilators, steroids, hospitalizations for respiratory causes

SECONDARY OUTCOMES:
Lung function parameters | 6 months of life
  Tidal volume (ml)
Lung function parameters 2 | 6 months of life
  Respiratory rate (breaths per minute)
Lung function parameters 3 | 6 months of life
  Time to peak expiratory flow/expiratory time (ratio)
Lung function parameters 4 | 12 months of life
  Functional residual capacity (ml)
Lung function parameters 5 | 12 months of life
  Lung clearance index 2.5 and 5.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Nobile, MD, PhD, MSc, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided